CLINICAL TRIAL: NCT06681766
Title: A Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneous Nomlabofusp in Adolescents and Children With Friedreich's Ataxia
Brief Title: A Study to Assess Nomlabofusp in Adolescents and Children With Friedreich's Ataxia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Review of Cohort 1 data facilitated direct enrollment into open label study and eliminate pause in study drug administration between PK study and open label study.
Sponsor: Larimar Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIN-1601-103
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nomlabofusp (Experimental): Subcutaneous injection of 0.8 mg/kg, with a maximum dose of 50 mg, once daily for 7 days
  Interventions: Drug: Nomlabofusp
- Placebo (Placebo Comparator): Subcutaneous injection once daily for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nomlabofusp — Nomlabofusp is a recombinant fusion protein provided in a sterile, preservative-free buffered solution for subcutaneous injection intended to deliver human frataxin, the protein deficient in Friedreich's ataxia.
  Other Names: CTI-1601
  Arms: Nomlabofusp
Drug: Placebo — The placebo is a sterile, preservative-free, clear liquid for subcutaneous injection.
  Other Names: CTI-1601 Placebo, Nomlabofusp Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the safety and tolerability of nomlabofusp (CTI-1601) in adolescents and children with Friedreich's ataxia (FRDA).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study evaluating a weight-based dose of nomlabofusp versus placebo in adolescents and children with FRDA. The study will consist of at least two cohorts with at least 12 to 15 participants in each cohort. Participants will be dosed once daily (QD) for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has genetically confirmed diagnosis of FRDA manifested by homozygous GAA repeat expansions, with repeat sizing (if available) included on the diagnosis report.
2. Male or female subjects ≥ 2 to < 18 years of age at screening.
3. Subjects must weigh ≥ 10.0 kg.
4. Subject must be able to traverse a distance of 25 feet with or without some assistive device (e.g., cane, walker, crutches, self-propelled wheelchair) and meet the following requirements:

   1. Be able to sit upright with thighs together and arms crossed without requiring support on more than 2 sides;
   2. Be able to transfer from bed to chair independently or with assistance if, in the opinion of the investigator, the degree of physical disability does not result in undue risk to the subject while participating in the study; and
   3. Perform basic age-appropriate daily care, such as feeding themselves and personal hygiene, with minimal assistance.

Exclusion Criteria:

1. Subjects who are confirmed as compound heterozygous (GAA repeat expansion on only 1 allele) for FRDA.
2. Subject has any condition, disease, or situation, including a cardiac condition or disease, that in the opinion of the investigator could confound the results of the study or put the subject at undue risk, making participation inadvisable.
3. Subjects currently receiving or having received omaveloxolone within 30 days prior to Screening.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Number of AEs, TEAEs, related TEAEs, Grade 3/4 TEAEs, and SAEs | Up to 72 days (including screening)
  Number
Number of subjects with ISRs | Up to 37 days
  Number
Change from baseline in electrocardiogram (ECG) parameter - heart rate (HR) | Baseline, Day 7
  Number
Change from baseline in electrocardiogram (ECG) parameter - PR interval | Baseline, Day 7
  Number
Change from baseline in electrocardiogram (ECG) parameter - QRS complex | Baseline, Day 7
  Number
Change from baseline in electrocardiogram (ECG) parameter - QT interval | Baseline, Day 7
  Number
Change from baseline in electrocardiogram (ECG) parameter - QTcF (Corrected QT Interval) | Baseline, Day 7
  Number
Change from baseline in echocardiogram (ECHO) parameter - ejection fraction (EF) | Baseline, Day 7
  Number
Change from baseline in echocardiogram (ECHO) parameter - left ventricular end-diastolic volume (LV EDV) | Baseline, Day 7
  Number
Change from baseline in echocardiogram (ECHO) parameter - left ventricular end-systolic volume (LV ESV) | Baseline, Day 7
  Number
Change from baseline in echocardiogram (ECHO) parameter - relative wall thickness (RWT) | Baseline, Day 7
  Number
Change from baseline in echocardiogram (ECHO) parameter - left ventricular mass (LVM) | Baseline, Day 7
  Number
Change from baseline in echocardiogram (ECHO) parameter - left ventricular posterior wall thickness | Baseline, Day 7
  Number
Change from baseline in echocardiogram (ECHO) parameter - septal wall thickness | Baseline, Day 7
  Number
Change from baseline in echocardiogram (ECHO) parameter - mitral valve inflow Doppler | Baseline, Day 7
  Number
Change from baseline in echocardiogram (ECHO) parameter - tissue Doppler | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - sodium | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - potassium | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - glucose | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - blood urea nitrogen | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - creatinine | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - calcium, chloride | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - phosphorus | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - total protein | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - total CO2 | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - albumin | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - AST | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - ALT | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - GGT | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - ALP | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - total bilirubin | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - uric acid | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - HbA1c | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - hemoglobin | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - hematocrit | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - RBC count | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - RDW | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - MCV | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - MCH | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - platelet count | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - WBC count | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - ANC | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - Eosinophils | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - Monocytes | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - Basophils | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - Lymphocytes | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - Bands | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - Neutrophils | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - Cholesterol | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - HDL cholesterol | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - LDL cholesterol | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - Triglycerides | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - very low-density lipoprotein cholesterol | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - pH | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - protein | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - blood | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - ketones | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - bilirubin | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - urobilinogen | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - nitrites | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - leukocyte esterase | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - color | Baseline, Day 7
  Number
Change from baseline in clinical laboratory assessment - specific gravity | Baseline, Day 7
  Number
Change from baseline in pulse rate | Baseline, Day 7
  Number
Number of subjects with abnormal physical examinations | Up to 72 days (including screening)
  Number
Number of subjects with suicidal ideation, suicidal behavior, and suicidal ideation or behavior based on the Columbia Suicide Severity Rating Scale (C-SSRS) | Up to 72 days (including screening)
  Number
Number of subjects who discontinue treatment and/or study | Up to 37 days
  Number

SECONDARY OUTCOMES:
AUC0-last | Days 1, 7
  Area under the concentration-time-curve to the last quantifiable timepoint
Cmax | Days 1, 7
  Maximum observed concentration
Tmax | Days 1, 7
  Time of maximum observed concentration
Ctrough | Days 1, 7
  Predose concentration
Change from baseline in FXN concentrations normalized to total protein observed in buccal cells collected from cheek swabs | Baseline, Day 7
  Number

CONTACTS AND LOCATIONS:
Overall Officials: Larimar Therapeutics, Inc., Study Chair — Larimar Therapeutics, Inc.
Locations (1):
- Uncommon Cures, Chevy Chase, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delatycki MB, Corben LA. Clinical features of Friedreich ataxia. J Child Neurol. 2012 Sep;27(9):1133-7. doi: 10.1177/0883073812448230. Epub 2012 Jun 29. PMID 22752493
- [Background] Deutsch EC, Santani AB, Perlman SL, Farmer JM, Stolle CA, Marusich MF, Lynch DR. A rapid, noninvasive immunoassay for frataxin: utility in assessment of Friedreich ataxia. Mol Genet Metab. 2010 Oct-Nov;101(2-3):238-45. doi: 10.1016/j.ymgme.2010.07.001. Epub 2010 Jul 8. PMID 20675166
- [Background] Fahey MC, Corben L, Collins V, Churchyard AJ, Delatycki MB. How is disease progress in Friedreich's ataxia best measured? A study of four rating scales. J Neurol Neurosurg Psychiatry. 2007 Apr;78(4):411-3. doi: 10.1136/jnnp.2006.096008. Epub 2006 Oct 20. PMID 17056635
- [Background] Goodkin DE, Hertsgaard D, Seminary J. Upper extremity function in multiple sclerosis: improving assessment sensitivity with box-and-block and nine-hole peg tests. Arch Phys Med Rehabil. 1988 Oct;69(10):850-4. PMID 3178453
- [Background] Indelicato E, Nachbauer W, Eigentler A, Amprosi M, Matteucci Gothe R, Giunti P, Mariotti C, Arpa J, Durr A, Klopstock T, Schols L, Giordano I, Burk K, Pandolfo M, Didszdun C, Schulz JB, Boesch S; EFACTS (European Friedreich's Ataxia Consortium for Translational Studies). Onset features and time to diagnosis in Friedreich's Ataxia. Orphanet J Rare Dis. 2020 Aug 3;15(1):198. doi: 10.1186/s13023-020-01475-9. PMID 32746884
- [Background] Koeppen AH. Friedreich's ataxia: pathology, pathogenesis, and molecular genetics. J Neurol Sci. 2011 Apr 15;303(1-2):1-12. doi: 10.1016/j.jns.2011.01.010. PMID 21315377
- [Background] Lawerman TF, Brandsma R, Burger H, Burgerhof JGM, Sival DA; the Childhood Ataxia and Cerebellar Group of the European Pediatric Neurology Society. Age-related reference values for the pediatric Scale for Assessment and Rating of Ataxia: a multicentre study. Dev Med Child Neurol. 2017 Oct;59(10):1077-1082. doi: 10.1111/dmcn.13507. Epub 2017 Aug 17. PMID 28815574
- [Background] Lazaropoulos M, Dong Y, Clark E, Greeley NR, Seyer LA, Brigatti KW, Christie C, Perlman SL, Wilmot GR, Gomez CM, Mathews KD, Yoon G, Zesiewicz T, Hoyle C, Subramony SH, Brocht AF, Farmer JM, Wilson RB, Deutsch EC, Lynch DR. Frataxin levels in peripheral tissue in Friedreich ataxia. Ann Clin Transl Neurol. 2015 Aug;2(8):831-42. doi: 10.1002/acn3.225. Epub 2015 Jul 1. PMID 26339677
- [Background] Pandolfo M. Friedreich ataxia. Arch Neurol. 2008 Oct;65(10):1296-303. doi: 10.1001/archneur.65.10.1296. PMID 18852343
- [Background] Rudick R, Antel J, Confavreux C, Cutter G, Ellison G, Fischer J, Lublin F, Miller A, Petkau J, Rao S, Reingold S, Syndulko K, Thompson A, Wallenberg J, Weinshenker B, Willoughby E. Clinical outcomes assessment in multiple sclerosis. Ann Neurol. 1996 Sep;40(3):469-79. doi: 10.1002/ana.410400321. PMID 8797541